CLINICAL TRIAL: NCT06150911
Title: A Study of Pain, Anxiety, and Impacts on Oral Health-related Quality of Life(OHRQoL) for Patients Before, During and After Orthodontic Treatment
Brief Title: Pain, Anxiety, and Impacts on Oral Health-related Quality of Life for Patients With Orthodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(II)-20230166
Record Dates: First submitted 2023-11-01; First posted 2023-11-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-07

CONDITIONS: Pain; Anxiety; Oral Health Related Quality of Life
Keywords: Visual Analogue Scale(VAS) pain scale; Generalized Anxiety Disorder 7-item (GAD-7) scale; Oral health impact profile-14(OHIP-14) scale
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about pain, anxiety, and impacts on oral health-related quality of life(OHRQoL) for patients before, during and after orthodontic treatment. The recruited participants with good health are from Kaohsiung medical university and local dental clinics .

The main questions it aims to answer are:

1. The differences of pain, anxiety, and impacts on oral health-related quality of life(OHRQoL) for patients before, during and after orthodontic treatment.
2. The correlation of pain, anxiety and oral health-related quality of life in our participant
3. The differences of seven domain in OHIP-14 scale in our participants The participants are asked to complete a self-administered in different time point.

DETAILED DESCRIPTION:
Orthodontic treatment is a common dental procedure aimed at improving teeth and bite alignment issues. Patients may experience various challenges before, during, and after orthodontic treatment, including pain, anxiety, and the impact on oral health-related quality of life. Here are some aspects to consider in researching these areas:

Pain: Orthodontic treatment typically causes a certain level of discomfort and pain. Research can focus on assessing changes in the intensity and frequency of pain experienced by patients before, during, and after treatment. Pain can be evaluated using visual analog scales or numerical rating scales, and the duration and relief of pain should be tracked.

Anxiety: Orthodontic treatment may induce anxiety and stress in some patients. Studies can assess anxiety levels at different stages of treatment through surveys or psychological measurement tools like anxiety assessment scales. Additionally, observing patients' behavior and emotional responses during treatment can provide insights into their anxiety levels.

Oral Health-Related Quality of Life: The success of orthodontic treatment is not solely determined by tooth movement but also relates to patients' oral health-related quality of life indicators. These indicators may include oral hygiene habits, dietary changes, and satisfaction with the treatment process. Questionnaires, oral examinations, and oral health-related quality of life assessment tools can be used to evaluate these aspects.

Researching these areas can help us gain a better understanding of patients' experiences and needs during orthodontic treatment. This, in turn, can aid in improving treatment methods and providing better patient care. Furthermore, research findings can be used to offer education and guidance to patients before, during, and after treatment to alleviate their pain and anxiety and promote oral health maintenance.

In summary, orthodontic treatment can significantly benefit patients in terms of addressing bite alignment issues and improving their psychological, physiological, and social interactions. However, in Taiwan, there is a lack of systematic research on the changes in pain, anxiety, and oral health-related quality of life indicators experienced by patients before, during, and after orthodontic treatment. Therefore, this study aims to investigate these issues through structured questionnaires among patients undergoing orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patient with clinical diagnosis malocclusion
* Age from 18 to 60 years old

Exclusion Criteria:

* Systemic and psychological disease
* Craniofacial deformity
* Received orthodontic treatment beforehand

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Study Population: study population are orthodontic patients which are recruited from orthodontic department ,Kaohsiung medical university and local dental clinics
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) pain scale | 2 years
  The pain scale illustrate the pain level which ranging from 0~10. 0 represent no pain,and 10 represent the most painful sensation. The participant will choose the most suitable pain sensation during the testing time point.
Generalized Anxiety Disorder 7-item (GAD-7) scale | 2 years
  The GAD-7 scale using seven questions to test the anxiety level measurement caused by any problems, and how difficult have these problems interfere you to do your work, take care of things at home, or get along with other people? Each question is measured with four point Likert's scale from 0~3 and then sum up to have the total score. The total score ranging from 0~4: extreme mild anxiety / 5~9: mild anxiety/ 10~14:moderate anxiety/15~21: severe anxiety.
Oral health impact profile(OHIP)-14 scale; self-administered questionnaire | 2 years
  The OHIP-14 scale was used to measure the participants' oral health related quality of life and it has seven conceptualized domains (two items per domain): functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap.In which, respondents are asked to rate how frequently they experienced an oral health impact (as described by each item). In turn, the response to each item is scored on a five-point Likert scale: 0, never; 1, hardly ever; 2, occasionally; 3, fairly often; and 4, very often or every day. Thus, summary OHIP-14 scores can range from 0 to 56. A high total value indicates a high negative impact on the OHRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Tseng, PHD, Study Chair — Kaohsiung Medical University
Locations (1):
- Kaohsiung medical university, Kaohsiung City, Taiwan